CLINICAL TRIAL: NCT06454461
Title: Efficacy of Upadacitinib After Autologous Non-cultured Epidermal Cell Suspension Transplantation in Vitiligo Participants -- a Pilot, Random, Observer Blinded, Comparative Study
Brief Title: Efficacy of Upadacitinib After NECS in Vitiligo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Shanshan Li, Dr., Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLi
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-08

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Experimental): upadacitinib after autologous non-cultured epidermal cell suspension transplantation
  Interventions: Drug: Upadacitinib 15 MG
- B (No Intervention): autologous non-cultured epidermal cell suspension transplantation

INTERVENTIONS:
Drug: Upadacitinib 15 MG — Upadacinib 15mg once daily for the 8 weeks after NECS
  Other Names: NECS
  Arms: A

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of upadacitinib after NECS in participants with vitiligo. The main question it aims to answer is: whether the short time use of upadacitinib after NECS will improve NECS efficacy. Participants in the experimental group will receive upadacitinib after NECS, while Participants in the control group will receive NECS only.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who can sign the informed consent.
2. Participants aged 18-60 years (both men and women) at the time of signing the informed consent.
3. Non-segmented vitiligo
4. Vitiligo affected area should meet the following two criteria:

(1) containing the target area (relatively flat vitiligo lesions except of the hands and feet, perineum, lips, joints, perianal); (2) total BSA involvement ≤30% 5. Clinically stable for more than one year (stable refers to the original lesion no longer expanding and no new lesions appearing).

6. All fertile women had to be willing to use at least one highly effective method of contraception from the time they signed informed consent through the final follow-up visit.

7. Participants must be willing and able to adhere to scheduled visits and scheduled treatments, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Any active skin lesions (e.g. psoriasis, dermatitis, skin ulceration, etc.) or skin infections (bacterial, fungal, viral, etc.) which may interfere with the assessment of vitiligo at screening.
2. Participants had a clinically significant infection (requiring hospitalization and parenteral treatment with antibiotics, antiviral agents, or antifungal agents for more than 3 days) within one month of the screening period or an active infection for which they were receiving treatment during the screening period.
3. Infected with HBV or HCV or HIV or syphilis.
4. Participants had active Tuberculosis or were receiving anti-Tuberculosis treatment, or had received anti-Tuberculosis treatment within 1 year.
5. Hepatic dysfunction (Total bilirubin ≥ 2 × ULN, AST≥2 × ULN, ALT ≥ 2 × ULN) at screening.
6. Renal impairment ( eGFR of <45 mL/min or receiving dialysis) at screening
7. Participants with malignancy or with a history of malignancy other than adequately treated or resected nonmetastatic basal cell carcinoma or squamous cell carcinoma.
8. Participants with current thyroid disease or undergoing thyroid replacement therapy.
9. Participants with a history of mental illness, such as anxiety or depression, who were assessed by the investigator to be unfit to participate in the study.
10. Pregnant or lactating female participants.
11. Participants who received any laser or phototherapy for vitiligo within 4 weeks before baseline.
12. Participants who received oral or systemic medications (e.g., glucocorticoids, cyclosporine, methotrexate, tacrolimus, Chinese medicine, etc.) aimed at controlling/improving vitiligo symptoms within 4 weeks before baseline.
13. Participants who had received JAK inhibitor therapy (including, but not limited to Ruxolitinib, Tofacitinib, Baricitinib, Upadacinib, etc.) within 12 weeks or 5 half-lives before baseline, whichever was longer.
14. Participants who had used any biologic agent within 12 weeks or 5 half-lives before baseline, whichever was longer.
15. Participants who had been enrolled in another intervention clinical trial within 4 weeks before the baseline visit or who were within 5 half-lives of the last dose of the intervention drug at baseline.
16. Any other condition that the investigator considered might render the subject ineligible for inclusion in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
T-VASI | 6 months
  Percentage of change from baseline in target lesion Vitiligo Area Scoring Index (T-VASI) at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology and Venerology, The First Hospital of Jilin University, No. 1 Xinmin Street, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
SCI articles published after the end of the trial can be shared with other researchers